CLINICAL TRIAL: NCT06300931
Title: Knowledge, Attitudes and Professional Behavior Towards Use of Silver Diamine Fluoride Among Dental Interns Before Versus After Educational Intervention.
Brief Title: KAP for Use of SDF Among Dental Interns Before vs After Educational Intervention
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mirette Yehia Ezzeldin Elwakil, Principal Investigator, Cairo University
Other Study IDs: KAPSDFE0948
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: SDF

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intern dentists: Group of interns to take KAP survey followed by a lecture and then another KAP survey
  Interventions: Other: educational lecture

INTERVENTIONS:
Other: educational lecture — An Educational lecture about SDF

SUMMARY:
This study is a KAP questionnaire to assess Egyptian intern dentists' knowledge, attitudes and practices regarding use of SDF before and after an educational intervention.

DETAILED DESCRIPTION:
The questionnaires will be distributed and filled out under the supervision of the primary investigator.

Each intern will be allowed to fill out the questionnaire. An educational lecture about SDF will follow. The questionnaires will be distributed and filled under the supervision of the primary investigator again.

ELIGIBILITY:
Inclusion Criteria:

Dental Interns who are enrolled in the pediatric dental department, Faculty of Dentistry, Cairo University who are willing to participate.

Exclusion Criteria:

Dental Interns who are enrolled in the pediatric dental department , Faculty of Dentistry, Cairo University who are unwilling to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Interns who graduated dental school and are currently enrolled in the pediatric dental department, Faculty of Dentistry, Cairo University
Sampling Method: Probability Sample
Enrollment: 638 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of knowledge levels and attitude regarding SDF use before educational intervention | 2 month
  A structured and validated questionnaire consisting of closed ended questions. Questionnaire used previously in a study done by Antonioni, Mario, et al., (2019) The questionnaire will be constructed in English

SECONDARY OUTCOMES:
Assessment of knowledge levels and attitude regarding SDF use after educational intervention Correlation between demographic data and use of SDF. | 2 month
  A structured and validated questionnaire consisting of closed ended questions. Questionnaire used previously in a study done by Antonioni, Mario, et al., (2019) The questionnaire will be constructed in English

IPD SHARING:
Plan to Share IPD: No